CLINICAL TRIAL: NCT03979989
Title: An Open-Label, Two-Way Crossover, Drug-Interaction Study to Determine the Effect of Omeprazole on the Pharmacokinetics of an Immediate-Release Capsule of CG5503 in Healthy Subjects
Brief Title: Drug-drug Interaction Study to Evaluate the Effect of Omeprazole on CG5503 (Tapentadol)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Collaborators: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HP5503/20; R331333-PAI-1009 (Other: Collaborator code)
Record Dates: First submitted 2019-06-06; First posted 2019-06-10 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Pharmacokinetic
MeSH Terms: interventions — Omeprazole

STUDY DESIGN:
Intervention Model Description: Participants were randomized to 1 of 2 treatment sequences (AB or BA). There was a washout of at least 7 days between the CG5503 administrations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tapentadol IR (Experimental): A single oral dose of tapentadol IR was administered in a fasted state (Treatment A).
  Interventions: Drug: Tapentadol IR capsule
- Omeprazole, Tapentadol IR (Experimental): Oral doses of omeprazole were administered once daily in a fasted state on 4 consecutive days (Days -3 to 1), plus 1 capsule of CG5503 IR administered 2 hours after the administration of omeprazole on Day 1 (Treatment B).
  Interventions: Drug: Tapentadol IR capsule; Drug: Omeprazole capsule

INTERVENTIONS:
Drug: Tapentadol IR capsule — Tapentadol IR capsule containing 93 mg tapentadol hydrochloride.
Drug: Omeprazole capsule — Omeprazole capsule containing 40 mg omeprazole.
  Arms: Omeprazole, Tapentadol IR

SUMMARY:
This was a single center, open-label, two-way crossover, drug-drug-interaction study to determine the effect of multiple dosing of omeprazole on 4 consecutive days on the pharmacokinetics of a single dose of an immediate-release capsule of CG5503 (tapentadol) in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman, between 25 and 55 years of age, inclusive.
* Body mass index between 20 and 28 kg/square meter, inclusive, with a minimum body weight of 50 kg.
* Signed the informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.
* Women must be postmenopausal (no spontaneous menses for at least 2 years), surgically sterile, abstinent, or practicing or agree to practice an effective method of birth control if they are sexually active before entry and throughout the study (effective methods of birth control include prescription hormonal contraceptives, intrauterine devices, double-barrier method, and male partner sterilization). Women must have a negative serum beta-human chorionic gonadotropin pregnancy test at screening and a negative urine pregnancy test on Day -1 of Treatment Period 1.
* Healthy on the basis of pre-study physical examination, medical history, 12-lead electrocardiogram, vital signs, and clinical laboratory parameters (serum chemistry, serology, hematology, and urinalysis) performed within 21 days before administration of the first dose of study drug. NOTE: If the results of the chemistry, hematology, or urinalysis testing are not within the normal limits of the laboratory reference ranges, the participant may be included in the study only on the condition that the investigator judges the deviations not clinically relevant.
* Signed informed consent for pharmacogenomic testing indicating whether they do or do not wish to participate in the genetic part of the study. NOTE: Participation in the genetic testing component is not mandatory for participation in the study.
* Blood pressure (after the subject is supine for 5 minutes) between 100 and 140 mmHg systolic, inclusive, and 50 and 90 mmHg diastolic, inclusive.
* Are willing to follow the prohibitions and restrictions as specified in the protocol.

Exclusion Criteria:

* History of

  * seizure disorder or epilepsy, or
  * mild or moderate traumatic brain injury, stroke, transient ischemic attack, or brain neoplasm within 1 year of screening, or
  * severe traumatic brain injury (consisting of one or more of the following: brain contusion; intracranial hematoma; or episode(s) of more than 24 hours duration of unconsciousness or post-traumatic amnesia) within 15 years of screening, or
  * severe traumatic brain injury resulting in ongoing sequelae consisting of transient changes in consciousness or symptoms suggestive thereof at any time.
* History of clinically significant pulmonary, gastrointestinal, immunologic, endocrine, neurologic, psychiatric, thromboembolic disease or metabolic disturbances, or any current physical conditions that could interfere with the interpretation of the study results.
* History of clinically significant allergies, especially known hypersensitivity or intolerance to opioids, opioid antagonists (e.g., naloxone), benzodiazepines (e.g., diazepam, clonazepam, lorazepam), or any study drug formulation component or any of the excipients, or heparin (should the use of a heparin lock be necessary).
* Positive test for human immunodeficiency virus (HIV 1 and 2), hepatitis B, or hepatitis C.
* History of substance abuse or a positive test for drugs of abuse or alcohol at screening (including on the day before the initial administration of study drug in the first treatment period).
* Blood donation or acute loss of blood (more than 500 mL) during the 3 months before study drug administration or intention to donate blood or blood products during the study or within 1 month after the completion of the study.
* Women who are pregnant, or plan to become pregnant during the study, or who are breast-feeding.
* Participants for whom omeprazole treatment is contraindicated.
* Participants who have used or plan to use the following during the study:

  * prescription medication (except for birth control medications and hormone replacement therapy) within 14 days before the first study drug administration
  * monoamine-oxidase inhibitors (MAOIs) and serotonin-norepinephrine reuptake inhibitors (SNRIs) within 21 days before the first study drug administration
  * over-the-counter (OTC) medication, especially nonsteroidal anti-inflammatory drugs (NSAIDS) (e.g., ibuprofen) or herbal medication, within 14 days before the first study drug administration
  * alcohol, grapefruit, grapefruit juice, or Seville orange products within 48 hours before the first study drug administration.
* Have taken an investigational drug within the 30 days before study administration (Day 1) or within a period of less than 5 times the drug's half-life, whichever is longer.
* Plan to undergo surgery or other procedures during the course of the study.
* Consume alcohol in quantities greater than 3 drinks every day (1 drink is defined as 12 ounces [approximately 360 mL] of beer, 4 ounces [approximately 120 mL] of wine, or 1 ounce [approximately 30 mL] of hard liquor).
* Regularly smoke more than 10 cigarettes/day or the equivalent.
* Unable to refrain from smoking or limit intake of caffeine or methylxanthine-containing foods or beverages (including chocolate) for 2 hours before and for 24 hours after study drug administration in both treatment periods.
* Unable to swallow solid, oral dosage forms whole with the aid of water (participants may not chew, divide, dissolve, or crush the study drug).
* Employees of the investigator or study center, with direct involvement in the proposed study or other studies under the direction of the investigator or study center, and family members of the employees or the investigator.
* In the opinion of the investigator, are subjects who are not likely to complete the study for whatever reason or who have an inability to communicate meaningfully with the investigator and staff.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2005-09-28 (Actual); Primary Completion 2005-11-16 (Actual); Study Completion 2005-11-16 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter: Cmax of CG5503 base | Pre-dose up to 48 hours post-dose
  14 blood samples for the determination of serum concentrations were taken at pre-dose and up to 48 hours after administration of the CG5503 IR capsule. The evaluation of the maximum observed serum concentration (Cmax) was based on the CG5503 base concentrations measured in serum samples using a validated liquid chromatography/tandem mass spectrometry (LC-MS/MS) method.
Pharmacokinetic parameter: AUC0-t of CG5503 base | Pre-dose up to 48 hours post-dose
  14 blood samples for the determination of serum concentrations were taken at pre-dose and up to 48 hours after administration of the CG5503 IR capsule. The evaluation of the area under the concentration time curve (AUC) from 0 hours to time t (=48 hours) (AUC0-t) was based on the CG5503 base concentrations measured in serum samples.
Pharmacokinetic parameter: AUC0-inf of CG5503 base | Pre-dose up to 48 hours post-dose
  14 blood samples for the determination of serum concentrations were taken at pre-dose and up to 48 hours after administration of the CG5503 IR capsule. The AUC from 0 hours to infinity (AUC0-inf) was extrapolated from the AUC from administration to the last measured concentration.

SECONDARY OUTCOMES:
Pharmacokinetic parameter: Cmax of CG5503-O-glucuronide | Pre-dose up to 48 hours post-dose
  14 blood samples for the determination of serum concentrations were taken at pre-dose and up to 48 hours after administration of the CG5503 IR capsule. The evaluation of the maximum observed serum concentration (Cmax) was based on the CG5503-O-glucuronide concentrations measured in serum samples using a validated liquid chromatography/tandem mass spectrometry (LC-MS/MS) method.
Pharmacokinetic parameter: AUC0-t of CG5503-O-glucuronide | Pre-dose up to 48 hours post-dose
  14 blood samples for the determination of serum concentrations were taken at pre-dose and up to 48 hours after administration of the CG5503 IR capsule. The evaluation of the area under the concentration time curve (AUC) from 0 hours to time t (=48 hours) (AUC0-t) was based on the CG5503-O-glucuronide concentrations measured in serum samples.
Pharmacokinetic parameter: AUC0-inf of CG5503-O-glucuronide | Pre-dose up to 48 hours post-dose
  14 blood samples for the determination of serum concentrations were taken at pre-dose and up to 48 hours after administration of the CG5503 IR capsule. The AUC from 0 hours to infinity (AUC0-inf) was extrapolated from the AUC from administration to the last measured concentration.
Incidence of treatment emergent adverse events | Day 1 to Day 4
  Number of adverse events and number of participants with adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director Grünenthal, Study Director — Grünenthal GmbH
Locations (1):
- J&JPRD Clinical Pharmacology Unit, Merksem, Belgium

IPD SHARING:
Plan to Share IPD: No